CLINICAL TRIAL: NCT07100431
Title: Comparison of Safety and Clinical Effects of Straight and Articulated Instruments (ArtiSential) in Laparoscopic Gastrectomy for Gastric Cancer Patients, a Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2022-0165
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Gastric Adenocarcinoma Patients, Who Are Scheduled for Laparoscopic Radical Gastrectomy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: During supra-pancreatic lymph node dissection, the assistant provides downward traction on the pancreas head with an instrument in their left hand to secure a clear surgical view. In the Control group, a conventional straight laparoscopic instrument was used for this purpose, while in the Articulating group, an articulating laparoscopic instrument (ArtiSential®, LIVSMED, Maryland jaw) was used.
Masking Description: Patients were randomly assigned in a 1:1 ratio to two groups; the control group or the experimental (Articulating) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Articulating group (Experimental): During supra-pancreatic lymph node dissection, the assistant provides downward traction on the pancreas head with an articulating laparoscopic instrument (ArtiSential®, LIVSMED, Maryland jaw) in their left hand.
  Interventions: Procedure: Articulating (experimental group); Procedure: Control (control group)
- Control group (No Intervention): During supra-pancreatic lymph node dissection, the assistant provides downward traction on the pancreas head with a conventional straight laparoscopic instrument in their left hand.

INTERVENTIONS:
Procedure: Articulating (experimental group) — 1. Surgical procedure On the day of surgery, random allocation to either the experimental or the control group will be perfored just before the start of the procedure. All of the surgery will be conducted laparoscopically. The control group will undergo surgery using a conventional straight laparoscopic instrument, while the experimental group will use an articulating instrument. The surgical procedure will be the same for both groups. The total time of surgery and the time spent on the supra-pancreatic lymph node dissection will be recorded during the procedure. The estimated blood loss during surgery will be also measured.
  Arms: Articulating group
Procedure: Control (control group) — 2. Postoperative follow-up Patients participating in this study will have the same postoperative care as those not participating in this study. To compare the degree of pancreatic injury, amylase and lipase levels will be measured in the serum and the peritoneal fluid frome the drainage on postoperative days 1 and 3.
  Postoperative complications will be classified and recorded according to the Clavien-Dindo classification for all complications occurring within 30 days after surgery. The dissected lymph nodes will be categorized by region, and the number of dissected lymph nodes will also be confirmed.
  Arms: Articulating group

SUMMARY:
In patients with gastric cancer, gastrectomy can be performed via laparoscopic/robotic or open surgery. It is crucial to completely remove the tumor along with an adequate extent of lymph node dissection. The number of lymph nodes retrieved during gastrectomy is considered an important factor associated with the quality of the surgery and can serve as an indicator of the completeness of the procedure.

In particular, during the dissection of lymph node stations 8, 9, 11p and 12a - which are located near the superior aspect of the pancreas - pressure is often applied to the pancreas to secure an adequate surgical view. Recent studies have suggested that this may be associated with postoperative pancreatic complications.

It is believed that the use of articulating instruments during laparoscopic gastrectomy may enable a safer dissection of lymph nodes located above the pancreas. However, to date, there have been lack of studies comparing the safety and efficacy of articulating versus straight instruments in laparoscopic gastrectomy. Therefore, this study aims to analyze the compare these two approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with gastric adenocarcinoma pathologically before surgery
2. Patients scheduled for laparoscopic radical gastrectomy
3. Patients aged more than 20
4. Patients with an ECOG 0 or 1

Exclusion Criteria:

1. Patients with a history of gastrectomy
2. Patients with a history of pancreatitis or pancreatic surgery
3. Patients with a history of abdominal surgery who are expected to have severe intra-abdominal adhesions
4. Patients scheduled for total gastrectomy with D2 lymph node dissection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The reduction in operative time achieved by using an articulating instrument for dissection of suprapancreatic lymph nodes during laparoscopic gastrectomy | During surgery, the total operation time, and the supra-pancreatic lymph node dissection time will be calculated respectively. The supra-pancreatic lymph node dissection time will be measured from the point of right gastric artery ligation to just before
  To confirm that the use of articulating instruments in radical gastrectomy can lead to more efficient and safer surgery compared to conventional straight instruments.

SECONDARY OUTCOMES:
The degree of pancreas injury after surgery | Amylase levels will be measured in serum and peritoneal fluid on postoperative day 1 and 3.
  To confirm that the use of articulating instruments in radical gastrectomy can lead to more efficient and safer surgery compared to conventional straight instruments.
Estimated blood loss | Estimated blood loss will be calculated during surgery.
  To confirm that the use of articulating instruments in radical gastrectomy can lead to more efficient and safer surgery compared to conventional straight instruments.
The number of retrieved lymph nodes | The number of retrieved lymph nodes were counted after surgery
  To confirm that the use of articulating instruments in radical gastrectomy can lead to more efficient and safer surgery compared to conventional straight instruments.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided